CLINICAL TRIAL: NCT02220673
Title: Serial Lung Function Measurements in 12 Healthy and 48 Mild Asthmatic Adults After Oral Inhalation of Ethanolic Solutions Containing Two Concentrations of the Excipient Butylated Hydroxytoluene (BHT, 0.1% and 0.5%) Administered With the Respimat® B (RMT-B) vs. Corresponding RMT-B and HFA MDI Without BHT; Repeated Increasing Doses With 2, 4, and 6 Actuations of Low Concentration Prior to High Concentration on Separate Days, Double Blind for RMT-B Use, Randomised 4-way Cross-over Design
Brief Title: Serial Lung Function Measurements in Healthy and Mild Asthmatic Adults After Oral Inhalation of Ethanolic Solutions Containing Two Concentrations of the Excipient Butylated Hydroxytoluene (BHT) Administered With the Respimat® B (RMT-B)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1256.13
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

ARMS (4):
- BHT 0.1% (Experimental)
  Interventions: Drug: BHT 0.1%
- BHT 0.5% (Experimental)
  Interventions: Drug: BHT 0.5%
- Placebo for RMT-B (Placebo Comparator)
  Interventions: Drug: Placebo for RMT-B
- Placebo for HFA-MDI (Placebo Comparator)
  Interventions: Drug: Placebo for HFA-MDI

INTERVENTIONS:
Drug: BHT 0.1%
  Arms: BHT 0.1%
Drug: BHT 0.5%
  Arms: BHT 0.5%
Drug: Placebo for RMT-B
  Arms: Placebo for RMT-B
Drug: Placebo for HFA-MDI
  Arms: Placebo for HFA-MDI

SUMMARY:
Primary objective: To investigate the safety and local tolerability of increasing cumulative doses (2, 4, 6 actuations) of a low (0.1%) and a high (0.5%) concentration of BHT administered via oral inhalation with the Respimat® inhaler B (RMT-B) vs. 2 inhalation solutions without BHT (placebo to BHT given by RMT B and placebo given by hydroxylfluoralkane metered dose inhaler (HFA MDI)). In a first step, the trial was performed in healthy subjects and - if no safety concerns arose - in a second step in patients with mild asthma who were sensitive to metacholine in a respective challenge test. Secondary objective: To explore the pharmacokinetics (PK) of BHT.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects

* Male or female adult subjects
* Age ≥ 18 and ≤ 65 years
* Body mass index (BMI) ≥ 18.5 and ≤ 32.0 kg/m2
* Non-smokers (within the last 5 years)
* Signed and dated written informed consent prior to admission to the trial in accordance with Good Clinical Practice (GCP) and the local legislation
* Proper use of RMT and MDI
* Able to perform technically satisfactory pulmonary function test

Patients with mild asthma

* Male or female adult subjects with intermittent and mild persistent asthma
* Age ≥ 18 and ≤ 65 years
* Body mass index (BMI) ≥ 18.5 and ≤ 32.0 kg/m2
* FEV1 ≥ 70% predicted and stable for at least 7 days prior to randomization
* Short acting beta agonist (SABA) response documented in the last 6 months
* A history of wheeze, cough, dyspnoea or chest tightness following exposure to at least one of the following: cold, exercise, dry air, smoke, dust, allergens
* Positive methacholine challenge test reflecting mild to moderate bronchial hyperreactivity (PC20: 0.25-4.0 mg/mL) performed within two weeks prior randomization (at visit 1 or between visit 1 and 2)
* None or stable dosages of pulmonary medications (SABA only) in the past 6 weeks
* Non smokers or ex-smokers for the last 5 years
* Signed and dated written informed consent prior to admission to the trial in accordance with GCP and the local legislation
* Proper use of RMT and MDI
* Able to perform technically satisfactory pulmonary function test

Exclusion Criteria:

Healthy subjects

* Any finding in the medical examination (including blood pressure (BP), pulse rate (PR)) deviating from normal and of clinical relevance
* Any laboratory value outside the reference range deemed of clinical relevance
* Pregnant or breast feeding women or women of childbearing potential without having a negative Human choriongonadotropin, β-subunit (ß-HCG) pregnancy test and without using a medically approved highly effective method of contraception for the previous 3 months
* Abnormal spirometry i.e., FEV1 <80% predicted and/or methacholine challenge at screening Visit 1 (or between Visits 1 and 2)
* Acute or chronic bacterial and viral infections of the lung
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Clinically relevant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Clinically relevant diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Use of drugs which might reasonably influence the results of the trial within 10 days prior to first administration or during the trial (assessed and judged by the investigator)
* Participation in another trial with an investigational drug within 1 month prior to administration or during the trial
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (>120 mL within 4 weeks prior to administration or during the trial)
* Excessive physical activities (within 1 week prior to administration or during the trial)
* Any vulnerable subjects
* Inability to comply with protocol requirements, instructions and study related restrictions, dietary regimen of trial site, and improbability of completing the study

Patients with mild asthma

* Any finding of the medical examination (including BP, PR) deviating from normal and of clinical relevance
* Any laboratory value that was of clinical relevance
* Moderate or severe persistent asthma
* Pregnant or breast feeding women or women of childbearing potential without a negative ß-HCG pregnancy test and without using a medically approved highly effective method of contraception for the previous 3 months
* Clinically relevant gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Clinically relevant diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* Chronic or relevant acute infections
* Treated or non-treated bacterial and viral infections of the lung, including active or latent tuberculosis
* Use of any corticosteroids, long acting muscarinic antagonist (LAMA) or long acting beta agonists (LABA), all within 1 month prior to screening Visit 1 and prior to administration of investigational product (i.e., allergic patients could only participate outside their season)
* Clinically relevant perennial allergies (i.e., which need actual treatment)
* Methylxanthines, antihistamines, antileukotrienes, cromolyn/nedocromil sodium all within 1 month prior to screening Visit 1 and prior to administration of investigational product
* SABAs 12 h prior to each visit day
* Use of other drugs which reasonably influence the results of the trial within 10 days prior to first administration or during the trial (e.g., beta blockers, all antimuscarinic agents like phenothiazines and some antidepressants)
* Participation in another trial with an investigational product within 1 month prior to administration or during the trial
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (>120 mL within 4 weeks prior to administration or during the trial)
* Excessive physical activities (within 3 days prior to administration or during the trial)
* Inability to comply with protocol requirements, instructions and trial related restrictions, dietary regimen of trial site, and improbability of completing the trial
* Any vulnerable patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Maximum decrease of forced expiratory volume in one second (FEV1) | baseline, 3 h after administration
  (Minimum FEV1 value over the interval 5 min to 2 h 50 min) minus (baseline value)

SECONDARY OUTCOMES:
Maximum decrease in FEV1 after 2 actuations | baseline, up to 50 minutes after drug administration
  (minimum FEV1 value over the interval 5 min to 50 min) - (baseline value)
Maximum decrease in FEV1 after 4 actuations | baseline, up to 1:50 hours after drug administration
  (minimum FEV1 value over the interval 1 h 5 min to 1 h 50 min) - (baseline value)
Maximum decrease in FEV1 after 6 actuations | baseline, up to 2:50 hours after drug administration
  (minimum FEV1 value over the interval 2 h 5 min to 2 h 50 min) - (baseline value)
Number of subjects with a decrease in FEV1 | baseline, up to 2:50 hours after drug administration
  stratified into classes of 0-20%, >20-40%, and >40%
Number of patients with cough episodes | up to 9 days
  within 5 min prior to the 1st inhalation and within 5 min after each of the 3 inhalations on each treatment day
Number of patients requiring rescue medication | up to 60 min after each dosing
Number of patients with adverse events | up to 10 days after the last treatment day
Cmax (maximum measured concentration of the analyte in plasma) | pre-dose, 2, 10, 25 and 55 min after each dosing
tmax (time from dosing to maximum measured concentration of the analyte in plasma) | pre-dose, 2, 10, 25 and 55 min after each dosing
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable concentration at tz) | pre-dose, 2, 10, 25 and 55 min after each dosing
Area under the curve (AUC) of FEV1 | over 3 hours after first dosing
AUC of FEV1 | over 1 hours after each dosing